CLINICAL TRIAL: NCT02646098
Title: CD34+ Selected Versus Unselected Autologous Stem Cell Transplantation in Advanced Stage Mantle Cell and Diffuse Large B-cell Lymphoma Patients, a Randomized Phase II Study
Brief Title: CD34+ Selected ASCT for Aggressive Lymphomas
Acronym: SAAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAAL-trial
Record Dates: First submitted 2015-11-04; First posted 2016-01-05 (Estimated); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Malignant Non-Hodgkin Lymphomas
Keywords: NHL; mantle cell lymphoma; diffuse large B-cell lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CD34+ cell selection (Active Comparator): CD34+ cell selection applying CliniMACS device (Miltenyi Biotec, Bergisch Gladbach, Germany)
  Interventions: Procedure: CD34+ cell selection
- No CD34+ cell selection (No Intervention): No CD34+ cell selection

INTERVENTIONS:
Procedure: CD34+ cell selection — CD34+ cell selection applying a CliniMACS device (Miltenyi Biotec, Bergisch Gladbach, Germany). This method for CD34+ cell selection will be used in this study and is considered as the standard treatment.
  Other Names: CD34+ selection
  Arms: CD34+ cell selection

SUMMARY:
Primary objective:

To assess the differences in the overall survival at 3 years of a CD34+ cell selection versus no selection of hematopoietic progenitor cells harvested during peripheral blood stem cell collection before high-dose chemotherapy with autologous stem cell transplantation (ASCT) in advanced stage mantle cell lymphoma (MCL) or diffuse large B-cell lymphoma (DLBCL) patients.

Secondary objectives:

To assess differences in disease-free survival between CD34+ cell selection versus no selection of hematopoietic progenitor cells harvested during peripheral blood stem cell collection before high-dose chemotherapy with autologous stem cell transplantation (ASCT) in advanced stage mantle cell (MCL) or in diffuse large B-cell lymphoma (DLBCL) patients.

To compare hematologic engraftment and the time needed until hematologic recovery after ASCT using CD34+ selected or unselected autologous stem cell grafts.

To compare infectious complications, particularly CMV infections, observed until 100 days after ASCT comparing CD34+ selected or unselected autologous stem cell grafts.

To assess the response rate at day 100 after ASCT in advanced stage mantle cell lymphoma (MCL) or diffuse large B-cell lymphoma (DLBCL) patients after ASCT comparing patients with CD34+ cell selection versus no selection.

To assess the total time needed for the apheresis procedure and the number of apheresis days needed to ensure the collection of a sufficient number of autologous stem cells comparing patients with CD34+ cell selection versus no selection.

To assess the need for the additional use of G-CSF (Neupogen) and of the stem cell releasing compound Plerixafor (Mozobil) to ensure the collection of a sufficient number of autologous stem cells comparing patients with CD34+ cell selection versus no selection.

Outcome(s):

The aim of the study is to show ≥ 15% better 3-year overall survival of lymphoma patients having received CD34+ cell selection during autologous stem cell collection before autologous stem cell transplantation compared to no CD34+ cell selection.

DETAILED DESCRIPTION:
Background and rationale: Autologous stem cell transplantation (ASCT): High-dose chemotherapy (HDCT) followed by ASCT is considered the treatment of choice for relapsed/refractory lymphomas. On the basis of the results of the PARMA study group trial, high-dose chemotherapy followed by ASCT has become the standard of care for patients with relapsed, chemo-sensitive aggressive lymphoma , and it is the treatment of choice in patients relapsing with diffuse large B-cell lymphomas (DLBCL), mantle cell lymphomas (MCL), follicular lymphoma (FL) or Hodgkin's disease (HD). Worldwide, about 11'000 patients are treated with ASCT per year because of relapsing lymphoma. The BEAM chemotherapy regimen is the most frequently used conditioning regimen before ASCT since more than thirty years.

Although HDCT with ASCT is a curative strategy for some patients with aggressive non-Hodgkin lymphoma (NHL), relapse or progression after ASCT is the major limitation of this procedure. Together with previously described factors that affect outcome after ASCT - such as prognostic score index, clinical response to induction or salvage chemotherapy, and the number of chemotherapy regimens received before ASCT - graft contamination with residual lymphoma cells is a major factor for disease relapse.

Graft contamination: Contamination of autologous graft by residual lymphoma cells has been demonstrated using several techniques including flow cytometry, immunohistochemistry or molecular methods. Subsequent studies have suggested that contamination with lymphoma cells contributes to relapse after ASCT using mobilized stem cells. A better outcome in syngenic transplantation in NHL compared with ASCT suggested the potential clinical benefit of purging the stem cell graft used for SCT.

Graft purging: The strategies implemented to remove lymphoma cells from harvested peripheral stem cells include complement-mediated use of lymphoma-directed antibodies, immunomagnetic beads, immunotoxins, or chemotherapeutic agents, as well as oncolytic viruses. Among them, CD34+ cell selection is an alternative and theoretically attractive strategy for tumor cell removal in lymphomas that do not express the CD34+ antigen. Various technologies have been used for positive selection of CD34+ cells, including immunomagnetic bead separation, avidin-biotin immunoaffinity systems, fluorescence-activated cell sorting, and magnetic-activated cell sorting (MACS). The feasibility and safety of CD34+ purified progenitor cell reinfusion after high-dose chemotherapy have also been demonstrated.

Clinical use of purged autologous grafts: Despite the theoretical advantage of using a purged graft in the ASCT setting, the standard procedure for ASCT involves the use of non-selected grafts. Whether the use of ex vivo purged grafts with CD34+ cell selection translates into improved long-term treatment outcome remains controversial. Noteworthy, not a single randomized study has been reported so far directly comparing in a prospective manner purged and unpurged grafts in ASCT. Thus, a randomized prospective direct comparison between these two procedures is long awaited and an unmet clinical need with presumably immediate impact on daily practice of ASCT.

Own experience with purged grafts: the investigator's institution has a long-standing experience with CD34+ cell selection applying the CliniMACS device (Miltenyi Biotec, Bergisch Gladbach, Germany). The investigator recently summarized the data in a retrospective analysis of advanced stage lymphoma patients comparing 31 patients with CD34+ cell selection versus 31 patients without selection (including 32 MCL and 30 DLBCL patients). Remarkably, the investigator found that the 5-year OS for selected versus not selected ASCT patients was 87% and 53% (p=0.004), and the 5-year PFS was 62% and 38% (p=0.031), respectively. These retrospective data suggest that using selected autografts for ASCT in advanced stage MCL and DLBCL is associated with significantly longer OS and PFS without increased toxicity, infectious complications or impaired engraftment. Finally, the investigator propose that these data provide the rationale for initiating a prospective randomized study on the use of CD34+ cell selection of grafts used for ASCT in patients with advanced-stage aggressive lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Eligible are patients with advanced stage (stage III or IV) malignant lymphomas including mantle cell lymphoma (MCL) in first or second remission or patients with diffuse large B-cell lymphoma (DLBCL) in first or second remission planned to undergo subsequent consolidation with standard high-dose chemotherapy with autologous stem cell transplantation.
* Patients must be aged 18-75 years, and must have given voluntary written informed consent.
* Negative pregnancy test (urine or serum) within 14 days prior to registration for all women of childbearing potential. Patients of childbearing potential must implement adequate measures (hormonal treatment p.o. or i.m., intra uterine surgical devices, or latex condoms) to avoid pregnancy during study treatment and for additional 12 months. No pregnant or lactating patients are allowed.

Exclusion Criteria:

* Patients not fit for autologous stem cell transplantation (ASCT).
* Patients with other serious medical condition that interfere with the completion of treatment according to this protocol or that would impair tolerance to therapy or prolong hematological recovery. Noteworthy, patients with seropositivity for HIV or for Hepatitis B and C are not excluded from this study if they are otherwise considered fit for ASCT.
* Acute uncontrolled infection
* Relevant co-existing disease excluding a treatment according to protocol
* HCTCI > 10
* Previous or concurrent malignant disease with the exception of basalioma/spinalioma of the skin, early-stage cervix carcinoma, or early-stage prostate cancer.
* Lack of patient cooperation to allow study treatment as outlined in this protocol.
* Pregnant or lactating female patients.
* Major coagulopathy or bleeding disorder.
* Major surgery less than 30 days before start of treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Overall survival of lymphoma patients having received CD34+ cell selection during autologous stem cell collection before autologous stem cell transplantation compared to no CD34+ cell selection

SECONDARY OUTCOMES:
Disease-free survival | 3 years
Engraftment as the time needed until hematologic recovery after ASCT | 100 days after ASCT
  Hematologic engraftment after ASCT is defined as the first day of neutrophils rising above 0.5 G/l, and of platelets rising above 20 G/L in the absence of platelet transfusions in the previous 3 days
Infectious complications | 100 days after ASCT
  Infectious complications, particularly CMV infections
Response rate | 100 days after ASCT
Total time needed for the apheresis procedure | 100 days after ASCT
Number of apheresis days needed to ensure the collection of a sufficient number of autologous stem cells | 100 days after ASCT
Acute and late toxicity/adverse events as assessed according to the CTCAE 4.0 | 100 days after ASCT
Need for the additional use of G-CSF (Neupogen) | 100 days after ASCT
Need for the stem cell releasing compound Plerixafor (Mozobil) | 100 days after ASCT

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pabst, Prof, Study Chair — Department for Medical Oncology; University Hospital/Inselspital; Freiburgstrasse 10; 3010 Bern; Gabriela Baerlocher, Prof, Principal Investigator — Universitätsklinik für Hämatologie und Hämatologisches Zentrallabor, Universitätsspital/Inselspital, 3010 Bern
Locations (1):
- Department for Medical Oncology; University Hospital/Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes